CLINICAL TRIAL: NCT07323992
Title: Effect of Modified Cawthorne-Cooksey Exercises on Cervical Proprioception and Functional Outcomes in Patients With Cervical Radiculopathy
Brief Title: To Investigate the Effect of Modified Cawthorne-cooksey Exercises on Cervical Proprioception and Functional Outcomes in Patients With Cervical Radiculopathy. Fifty Four Patients With Cervical Radiculopathy From Both Sexes Will be Selected Randomly and Allocated Into Two Equal Groups.
Acronym: Cawthorne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German International University (Other)
Responsible Party: Principal Investigator, Ahmed Khairy Abdullah Hussein, Teaching Assistant of Physical Therapy, German International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/006093
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical radiculopathy; disc; cervical; radiculopathy; nerve; root; compression
MeSH Terms: conditions — Radiculopathy | interventions — Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cawthorne-Cooksey exercises (Experimental): Cawthorne-Cooksey exercises are one form of vestibular exercises under this training involving centers such as visual, proprioceptive, and vestibular activities. Cawthorne-Cooksey exercises, originally developed for vestibular rehabilitation, focus on eye-head-body coordination and postural adaptation. When adapted for cervical use, they may enhance neuromuscular control, improve cervical joint position sense, and promote motor learning. These exercises are made to compensate for the affected vestibular signals (which cause poor balance and coordination) by retraining the eye and body musculatures.
  Interventions: Other: Cawthorne-Cooksey exercises; Other: Therapeutic Ultrasound
- Therapeutic Ultrasound (Experimental): Therapeutic Ultrasound:
  The application of ultrasound therapy with patient prone lying position paravertebral in posterior aspect of neck. The Treatment parameter ( 1 MHZ, FR 100HZ , duty factor 75% , power intensity 1.5w/cm2 , continuous mode , treatment time 5 min ).
  Interventions: Other: Therapeutic Ultrasound

INTERVENTIONS:
Other: Cawthorne-Cooksey exercises — Cawthorne-Cooksey exercises are one form of vestibular exercises under this training involving centers such as visual, proprioceptive, and vestibular activities.
  Cawthorne-Cooksey exercises, originally developed for vestibular rehabilitation, focus on eye-head-body coordination and postural adaptation. When adapted for cervical use, they may enhance neuromuscular control, improve cervical joint position sense, and promote motor learning. These exercises are made to compensate for the affected vestibular signals (which cause poor balance and coordination) by retraining the eye and body musculatures.
  Arms: Cawthorne-Cooksey exercises
Other: Therapeutic Ultrasound — The application of ultrasound therapy with patient prone lying position paravertebral in posterior aspect of neck. The Treatment parameter ( 1 MHZ, FR 100HZ , duty factor 75% , power intensity 1.5w/cm2 , continuous mode , treatment time 5 min ).

SUMMARY:
To investigate the effect of cawthorne-cooksey exercises on cervical proprioception and functional outcomes in patients with cervical radiculopathy

DETAILED DESCRIPTION:
Fifty four patients with cervical radiculopathy from both sexes will be selected randomly outpatient clinic and allocated into two equal groups. The Control Group will receive the selected physical therapy program only (electrotherapy, manual therapy, strengthening exercises), study Group will receive the Cawthorne-Cooksey exercises program and the selected physical therapy program. Basic assumptions

It will be assumed that:

* All the patients will follow the instructions and the rehabilitation program that are given to them.
* The motivation and cooperation are the same for all patients
* The patients will exert their maximum efforts during the study.

Null Hypothesis:

It will be hypothesized that:

* There will be no significant effect of Cawthorne-Cooksey exercises on proprioception in patients with cervical radiculopathy.
* There will be no significant effect of Cawthorne-Cooksey exercises on functional outcomes in patients with cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages range from 30 to 45 years.
2. Both sexes
3. With mild to moderate cervical disability according to the neck disability index.
4. Unilateral cervical radiculopathy for more than 6 months.
5. Cervical radiculopathy due to disc prolapse (C5-C6) (C6-C7) mild to moderate or disc prolapse according to magnetic resonance image(MRI).
6. Complaining from vertigo at least for 3 months.
7. Normal body mass index (18.5 - 24.99Kg/m2).

Exclusion Criteria:

1. Any other musculoskeletal disorders of the spine or upper extremity
2. Patients with any other Neurological deficits, psychiatric disease Cervical myelopathy, Cognitive problems, vertebral fractures and previous history of spine or cervical surgery.
3. Clinical instability, recent trauma.
4. Structural abnormalities of the spine, osteoporosis, and spasmodic torticollis.
5. Inflammatory or other specific disorders of spine such as ankylosing spondylitis and rheumatoid arthritis

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Cervical Proprioception | From enrollment to the end of treatment at 8 weeks
  Measuring Neck Proprioception by cervical joint position error via overhead laser pointer :
  1. Laser pointer: will be fixed to the subject's head by a strap to determine the degree of error in the test .
  2. Target paper: typically, 40 cm in diameter that contains concentric circles in 1 cm increments, divided into 4 quadrants intersecting at zero .
  3. Chair: a stable chair with back support and positioned such that it will not move when the subject will move his/her head during the test.
  4. Colored stickers: will be used to determine the starting and the ending points of the laser.
  5. Ruler: to measure the distance between the start point and endpoint in each direction on the target paper.

CONTACTS AND LOCATIONS:
Locations (1):
- Pivot clinic, Cairo, Egypt